CLINICAL TRIAL: NCT06904898
Title: CONDUIT vs. PEEK Cages in Patients Undergoing Direct Lateral Interbody Fusion (DLIF): A Randomized, Prospective Trial
Brief Title: CONDUIT vs. PEEK Cages
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 844964
Record Dates: First submitted 2025-03-07; First posted 2025-04-01 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Lumbar Degenerative Disease

STUDY DESIGN:
Who Masked: Participant
Masking Description: The study participants will be randomized to either receiving Cougar LS/Syncage ALIF or CONDUIT LLIF/ALIF cage at the time of surgery. utilizing GraphPad QuickCalcs, which is a closed-source, free, online limited randomization software for allocating subjects to a number of groups, with repeated block defaults at one. It can also produce a shuffled list of numbers for each group. After randomization, each patient will undergo DLIF using the standard surgical technique.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Conduit (Other): Patients undergoing DLIf (transposons or anterior-to-psoas approach) will be randomized to PEEK cages + rhBMP-2 vs. CONDUIT cages to compare the clinical outcomes and determine the associated cost.
  Interventions: Device: Cougar LS/Syncage ALIF or CONDUIT LLIF/ALIF cage
- PEEK + rh-BMP-2 cage (Other): Patients undergoing DLIf (transposons or anterior-to-psoas approach) will be randomized to PEEK cages + rhBMP-2 vs. CONDUIT cages to compare the clinical outcomes and determine the associated cost.
  Interventions: Device: Cougar LS/Syncage ALIF or CONDUIT LLIF/ALIF cage

INTERVENTIONS:
Device: Cougar LS/Syncage ALIF or CONDUIT LLIF/ALIF cage — Comparison between cages to determine the effectiveness and cost related to the study procedures.

SUMMARY:
In this study, the Principal Investigator aim to compare the clinical and radiographic outcomes of patients with degenerative lumbar disease undergoing direct lateral interbody fusion (DLIF) using two different types of lateral interbody cages: PEEK cages combined with rhBMP-2 versus CONDUIT cages. This will be a randomized, prospective, open-label clinical trial. By examining these two groups, the PI hope to determine whether PEEK cages with rhBMP-2 and CONDUIT cages are equally effective for DLIF procedures. The findings from this study will help us optimize the surgical approach for future patients undergoing DLIF.

DETAILED DESCRIPTION:
Direct lateral interbody fusion (DLIF) is a powerful surgical tool in a spine surgeon's armamentarium to address lumbar spine pathology minimally invasively. It has been widely adopted amongst spine surgeons to gain access to the lumbar disc through a small incision on a patient's flank. Through a retroperitoneal approach, the surgeon can perform discectomy, prep end plates, and insert an interbody cage with a much longer (lateral-medial) and wider (anterior-posterior) footprint than posterior lumbar interbody fusion (PLIF). Using either transpsoas or anterior-to-psoas (ATP) technique, the surgeons are now able to address lumbar spine pathologies affecting L2 to S1 minimally invasively. Both approaches are acceptable and widely adopted amongst spine surgeons. There are many commercially available FDA-approved DLIF cages in market for spine surgeons to use. The cages made of polyetheretherketone (PEEK) and titanium are most commonly used. Many surgeons who use PEEK cages in DLIF supplement the construct with recombinant human bone morphogenic protein-2 (rhBMP-2) to achieve fusion. PEEK has an inert and hydrophobic property which does not induce osteogenesis. In-vitro studies demonstrate absence of bone formation through PEEK. By adding rhBMP-2, it may induce robust osteoinduction around PEEK, achieving fusion across disk space over time. On the other hand, porous titanium has all three properties: osteoconductivity, osteoinductivity, and osseointegration. This may create a more favorable environment for fusion, which obviates the need for rhBMP-2 supplementation. Both types of cages are approved for the study's indications and are routinely used in DLIF at Penn. The surgical staff is qualified to implant both devices.

Aside from the type of cage used, subjects' DLIF procedures will not be altered for the purposes of the study. There are no known differences in the risks and benefits of the two cages being studied. Cage choice in routine care is based on each individual surgeon's standard-of-care preference. As such, there is a possibility of the patient getting either of these cages placed, should they choose to not participate in the study.

ELIGIBILITY:
Inclusion Criteria:

* • Patients with one to two consecutive level lumbar degenerative disease from L2to S1, including Grade 1 (<25%) Spondylolisthesis

  * Patients undergoing direct lateral interbody fusion (transpsoas or anterior-to-psoas approach) for lumbar disease
  * Skeletally mature patients, aged 18 and older
  * Patients able to fully comply with the clinical protocol and adhere to the follow-up schedule and protocol requirements
  * Patients able to understand and sign the study-specific, IRB approved informed consent form

Exclusion Criteria:

* • Spondylolisthesis greater than Grade 1

  * Traumatic lumbar disease
  * Spinal Deformity

    * Coronal Cobb angle greater than 40 degrees
    * Severe sagittal imbalance
  * Existing fusion construct longer than 2 consecutive levels
  * Active infection - systemic or local
  * Tumor diagnosis
  * Untreated osteoporosis, defined as T Spine < -2.5 on DEXA scan
  * Active smoking habit
  * Current incarceration
  * Pregnancy
  * Involvement in an active spinal litigation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-03-13 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Clinical outcomes | 24 months
  Difference in fusion rates for patients who get the PEEK + rh-BMP-2 cage and those who get the CONDUIT cage.
ODI scores | 24 months
  The ODI is comprised of ten items with associated statements for the patient to select which reflect the patient's ability to manage their everyday life while dealing with their pain. Each of the ten items in the ODI has six statements from which patients are requested to select one. This allows scoring from 0-5 for each item. A maximum score of 50 is possible. The score obtained by individual patients can be multiplied by 2, and this will provide a percentage score

SECONDARY OUTCOMES:
Cost | 24 months
  Costs associated with the PEEK + rh-BMP-2 and CONDUIT cages will be assessed.

CONTACTS AND LOCATIONS:
Locations (1):
- Pennsylvania Hospital, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided